CLINICAL TRIAL: NCT05404737
Title: Interchangeability of Right Ventricle Longitudinal Shortening Fraction Measurements Performed by Trans-thoracic and Trans-esophageal Echocardiography in the Operating Room
Brief Title: Interchangeability of Right Ventricle Longitudinal Shortening in Echocardiography
Acronym: RVLSBO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2021_843_0056
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Right Ventricle; Speckle Tracking; Strains; Cardiac Surgery
Keywords: Right ventricle; speckle tracking; Strains; cardiac surgery
MeSH Terms: conditions — Sprains and Strains

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: transthoracic echocardiography (TTE) — In order to evaluate the interchangeability of RV-LSF, a TTE will be performed just after the placement of general anesthesia, when the patient is under mechanical ventilation
Other: transoesophageal echocardiography (TEE). — During cardiopulmonary bypass surgery patients is monitored by a TEE as recommended.

SUMMARY:
RV longitudinal shortening fraction (RV-SLF) is based on the analysis of the tricuspid annulus displacement (TAD) and can be performed in transthoracic (TTE) or transoesophageal echocardiography (TEE). Having an 2D-STE interchangeable parameter would allow accurate measurement of RV systolic function before, during and after cardiac surgery. However, to date, there are no data on the interchangeability of RV-LSF measurements performed in TTE and TEE.

The aim of the study is to evaluate the interchangeability of TTE and TEE measurements of RV-LSF during cardiopulmonary bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (>18 years)
* Patient hospitalized at the Amiens University Hospital for scheduled cardiac surgery under cardiopulmonary bypass.
* Information of the patient and collection of his non-opposition

Exclusion Criteria:

* Patient with a contraindication to the realization of TEE (gastric or mediastinal pathology)
* Patient with poor echogenicity on TEE not allowing evaluation of 2D-STE parameters of the right ventricle
* Patient with a rapid supraventricular rhythm disorder (HR > 100) at the time of TTE and/or TEE.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Variation of the RV-LSF (in %) between TTE and TEE | one day
  RV-LSF is : Right ventricular longitudinal shortening fraction. RV-LSF is an angle-independent and automatically calculated speckle-tracking parameter and reproducible parameter.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Beyls C, Huette P, Vangreveninge P, Leviel F, Daumin C, Ammar B, Touati G, Roger B, Caus T, Dupont H, Abou-Arab O, Momar D, Mahjoub Y. Interchangeability of right ventricular longitudinal shortening fraction assessed by transthoracic and transoesophageal echocardiography in the perioperative setting: A prospective study. Front Cardiovasc Med. 2022 Dec 23;9:1074956. doi: 10.3389/fcvm.2022.1074956. eCollection 2022. PMID 36620637